# **Cover Page for SAP**

| Sponsor name: | Novo Nordisk A/S |
|---|---|
| NCT number | NCT05723835 |
| Sponsor trial ID: | NN8640 - 4469 |
| Official title of study: | A study evaluating the safety and efficacy of once - weekly dosing of somapacitan in a basket study design in paediatric participants with short stature either born small for gestational age or with Turner syndrome, Noonan syndrome or idiopathic short stature |
| Document date* | 24-June-2022 |

<sup>\*</sup>Document date refers to the date on which the document was most recently updated.


Date: 24 June 2022 Novo Nordisk
Version: 1.0
Status: Final


## **Statistical Analysis Plan**

### **Protocol Title:**

A study evaluating the safety and efficacy of once-weekly dosing of somapacitan in a basket study design in paediatric participants with short stature either born small for gestational age or with Turner syndrome, Noonan syndrome or idiopathic short stature.

### **Short title:**

A research study looking at how safe somapacitan is and how well it works in children who need help to grow – REAL 9

**Substance: Somapacitan** 

# **Table of contents**

| T | able o | of contents | 2 |
|---|---|---|---|
| T | able o | of figures | 3 |
| | | of tables | |
| | | n History | |
| L | ist of | abbreviations | 6 |
| 1 | Intro | oduction | 8 |
| | 1.1 | Objectives, Endpoints, and Estimands | |
| | 1.2 | Study Design | 9 |
| 2 | Stati | istical Hypothesis | 11 |
| | 2.1 | Multiplicity Adjustment | 11 |
| 3 | Ana | lysis Sets | 12 |
| 4 | | istical Analyses | |
| 4 | 4.1 | General Considerations | |
| | 4.2 | Primary Endpoint/Estimand Analysis | |
| | 2 | 4.2.1 Definition of Endpoint | |
| | | 4.2.2 Main Analytical Approach | |
| | | 4.2.3 Sensitivity Analysis | |
| | | 4.2.4 Supplementary Analysis | |
| | 4.3 | Secondary Endpoints/Estimands Analysis | |
| | | 4.3.1 Confirmatory Secondary Endpoints | |
| | 4.4 | 4.3.2 Supportive Secondary Endpoints/Estimands | |
| | 4.4<br>4.5 | Exploratory Endpoints Analysis | |
| | 4.3 | Other Safety Analysis | |
| | | 4.5.2 Adverse Events | |
| | | 4.5.3 Additional Safety Assessments | |
| | 4.6 | Other Analysis | |
| | | 4.6.1 Other parameters | 16 |
| | | 4.6.2 Subgroup Analysis | |
| | 4.7 | Interim Analysis | 17 |
| | 4.8 | Changes to Protocol-planned Analysis | 18 |
| 5 | Sam | ple size determination | 19 |
| 6 | Suni | porting Documentation | 20 |
| • | 6.1 | Appendix 1: Definition and calculation of endpoints, assessments and derivations | |
| 7 | Rofo | erences | |
| 1 | IXCIC | / VII VO | 4 |

1.0

| Statistical Analysis Plan<br>Study ID: NN8640-4469 | CONFIDENTIAL | Date:<br>Version:<br>Status: | 1.0<br>Final | Novo Nordisk |
|---|---|---|---|---|
| | | Page: | 3 of 24 | |
| 3 | | Version: | 1.0 | |

# Table of figures

| | Page |
|-----------------------|------|
| Figure 1 Study design | 10 |

Statistical Analysis Plan
Study ID: NN8640-4469


Date: 24 June 2022
Version: 1.0
Status: Final


## **Table of tables**

| | Page |
|-------------------------------------------------|------|
| Table 1 Objectives and endpoints | 8 |
| Table 2 Supportive secondary efficacy endpoints | 14 |
| Table 3 Overview of other parameters | 17 |

Statistical Analysis Plan
Study ID: NN8640-4469


Date: 24 June 2022 Version: 1.0
Status: Final 

# **Version History**

This Statistical Analysis Plan (SAP) for study NN8640-4469 is based on the protocol version 3.0 dated 21 December 2022.

| SAP Version | Date | Change | Rationale |
|-------------|--------------|----------------|------------------|
| 1.0 | 24 June 2024 | Not Applicable | Original version |


Date: 24 June 2022 Novo Nordisk
Version: 1.0

Version: 1.0 Status: Final 

### List of abbreviations

AE adverse event

BMI body mass index

DPS data points set

FAS full analysis set

FPFV first patient first visit

GH growth hormone

GH-INJ-CTB Growth Hormone Injection - Child Treatment Burden

GH-PPO Growth Hormone Patient Preference Questionnaire

HV height velocity

IGF-1 insulin-like growth factor 1

IGFBP-3 insulin-like growth factor binding protein-3

IMP investigational medical product

ISS idiopathic short stature

IVSed end-diastolic interventricular septum thickness

LVIDed end-diastolic left ventricular internal diameter

LVIDes end-systolic left ventricular internal diameter

LVPWed end-diastolic left ventricular posterior wall thickness

MAP modelling analysis plan

MedDRA medical dictionary for regulatory activities

MPH midparental target height

NAH near adult height

NS Noonan syndrome

PAS participant analysis set

PD pharmacodynamic

PK pharmacokinetic

| Statistical Analysis Plan<br>Study ID: NN8640-4469 | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 24 June 2022 Nove<br>1.0<br>Final<br>7 of 24 | o Nordisk |
|---|---|---|---|---|
| SAP | Statistical Analysis Plan | | | |
| SAS | safety analysis set | | | |
| SDS | standard deviation score | | | |
| SGA | small for gestational age | | | |
| TS | Turner syndrome | | | |


Date: Version: Status: Page:

24 June 2022 Novo Nordisk 1.0 Final 8 of 24

#### Introduction 1

Primary analysis of the primary endpoint addressing the primary estimand was defined in protocol before first patient first visit (FPFV). There are no changes to the analysis described in the protocol.

This SAP is based on the protocol: A study evaluating the safety and efficacy of once-weekly dosing of somapacitan in a basket study design in paediatric participants with short stature either born small for gestational age or with Turner syndrome, Noonan syndrome or idiopathic short stature. REAL 9, version 3.0 (dated 21 December 2022). This SAP covers specification of statistical considerations and analyses for efficacy and safety data. SAP 1.0 was created post FPFV.

#### 1.1 Objectives, Endpoints, and Estimands

#### Table 1 Objectives and endpoints

| Ob | jectives | Endpoints | | |
|---|---|---|---|---|
| Primary | | Title | Time frame | Unit |
| | | Primary endpoint: | | |
| | weekly somapacitan in children,<br>either naïve or non-naïve to GH<br>treatment, within each of the four<br>indications: SGA, TS, NS or ISS. | Number of adverse events (AEs) | From baseline (week 0) to week 26 | Number of<br>AEs |
| Sec | condary | Title | Time frame | Unit |
| • | To evaluate the long-term safety | Secondary supportive safety e | ndpoint: | |
| | of once-weekly somapacitan in children, either naïve or non-naïve to GH treatment, within each of the four indications: SGA, TS, NS or ISS. | Number of adverse events (AEs) possibly or probably related to somapacitan | From baseline (week 0) to week 26 | Number of AEs |
| | | Number of adverse events (AEs) | From baseline (week 0) to week 156 | Number of<br>AEs |
| • | To evaluate the efficacy of once-<br>weekly somapacitan for in<br>children, either naïve or non-<br>naïve to GH treatment, within | Secondary supportive efficacy endpoints: | | |
| | | Height Velocity | From baseline (week 0) to week 26 | cm/year |
| | each of the four indications: SGA, TS, NS or ISS. | Change in Height SDS | From baseline (week 0) to week 26 | Score* |
| | | Change in Height Velocity<br>SDS | From baseline (week 0) to week 26 | Score* |
| | | Change in IGF-1 SDS | From baseline (week 0) to week 26 | Score* |
| | | Change in IGFBP-3 SDS | From baseline (week 0) to week 26 | Score* |
| • | To evaluate the steady state | Secondary supportive efficacy endpoint: | | |
| | pharmacokinetics of once-weekly<br>somapacitan in children, either<br>naïve or non-naïve to GH<br>treatment, within each of the four<br>indications: SGA, TS, NS or ISS. | Weekly average somapacitan concentration (C <sub>avg</sub> ) based on population PK analysis | From baseline (week 0) to week 26 | ng/ml |

| Statistical Analysis Plan | | Date: | 24 June 2022 Novo Nordisk |
|---|---|---|---|
| • | CONFIDENTIAL | Status: | Final |
| | | Page: | 9 of 24 |

<sup>\*</sup>Positive score indicates that the value is closer to or above the reference population compared to baseline.

#### **Primary estimand**

The primary clinical question of interest is: What is the incidence of AEs from baseline to week 26 in the four populations (SGA, TS, NS or ISS) in all patients while on treatment regardless of dose reduction?

For the primary objective, the same primary estimand is defined for each of the four populations (SGA, TS, NS or ISS) with 5 attributes:

- The treatment condition of interest is defined as somapacitan regardless of dose reduction
- The population targeted by the clinical question: The treatment effect will be assessed separately for each of the four populations (SGA, TS, NS or ISS)
- Endpoint: Number of adverse events from baseline to 26 weeks
- Remaining intercurrent events:
  - Treatment discontinuation for any reason: Participants data will be included up to 14 days after treatment discontinuation. Data collected 14 days after the intercurrent event will be regarded as not relevant for estimation of the treatment effect
  - o Dose reduction due to IGF-I or AE: Is addressed by the treatment condition of interest attribute

There are no remaining intercurrent events

• Population-level summary: Event rate per 100 patient years

Rationale for estimand: The primary estimand assesses the expected safety profile in relation to incidence of AEs for a future population (SGA, TS, NS or ISS) while on somapacitan treatment for 26 weeks, if no treatment discontinuation occurs for any reason.

#### **Secondary estimands**

The supportive secondary safety estimand regarding the incidence of AEs possibly or probably related to somapacitan from baseline up to week 26 of somapacitan treatment will be evaluated in a similar way as the primary endpoint including possibly or probably related to somapacitan in the endpoint attribute.

The supportive secondary safety estimand regarding the incidence of AEs from baseline to week 156 of somapacitan treatment will be evaluated in a similar way as the primary endpoint substituting 156 weeks for 26 weeks.

The supportive secondary efficacy estimands will be specified in Section 4.3.2.

#### 1.2 Study Design

This is an interventional, multi-national, multi-centre, open-labelled, uncontrolled phase 3 study with a basket design. The study is designed to evaluate safety and efficacy of once-weekly dosing of somapacitan 0.24 mg/kg/week during 26 weeks (main phase) in children with short stature in each of the indications SGA, TS, NS and ISS. The 26-week main phase will be followed by a 130-week extension phase with once-weekly dosing of somapacitan 0.24 mg/kg/week to evaluate long-term safety. Study participants will include children with SGA, TS (only females), NS and ISS.

Approximately 60 participants in total are planned to be screened and up to 50 participants in total are planned to be enrolled (planned treated) in this study. In total, at least 40 participants are planned to complete the study. All participants will receive somapacitan 0.24 mg/kg/week.

| Statistical Analysis Plan | | Date: | 24 June 2022 | Novo Nordisk |
|---|---|---|---|---|
| | CONFIDENTIAL | Status: | Final | |
| | | Page: | 10 of 24 | |

The total treatment duration for each participant is scheduled to be 3 years. The treatment period is followed by a safety follow-up period of 30 days.

The study consists of:

- an up to 3-week screening period for participants in the indications SGA and ISS
- an up to 6-week screening period for participants in the indications TS and NS
- a 26-week interventional main phase
- a 130-week interventional extension phase
- a 30-day follow-up period

Figure 1 Study design




Date: 24 June 2022 Novo Nordisk
Version: 1.0
Status: Final


# 2 Statistical Hypothesis

No hypotheses are planned to be tested in the study.

## 2.1 Multiplicity Adjustment

Not applicable.

## 3 Analysis Sets

The following participant analysis sets are defined within each sub-study:

| Participant analysis set (PAS) | Description |
|---|---|
| Full analysis set (FAS) | All participants assigned to study intervention. |
| Safety analysis set (SAS) | All participants who are exposed to study intervention. |

The full analysis set will be used to analyse endpoints related to the efficacy objectives and the safety analysis set will be used to analyse the endpoints and assessments related to safety.

For the efficacy analyses, participants will be included in the analyses according to the planned investigational intervention; whereas for safety analyses, participants will be included in the analyses according to the investigational intervention they actually received.

The following data points sets are defined:

| Defined data points set (DPS) | Description |
|---|---|
| In-study | All observations from assignment to study intervention date up until visit 7 or last study contact, whichever comes first. |
| On-treatment | All observed data from first study intervention and up until visit 7, last study contact, or 14 days after last administration, whichever comes first. |

The on-treatment data point sets represent data collected in the period in which a participant is considered exposed to IMP.

FAS and In-study are used to estimate the supportive secondary efficacy estimands for Height velocity, Change in Height SDS and Change in Height Velocity SDS.

FAS and On-treatment are used to present the supportive secondary efficacy estimands for Change in IGF-I SDS and Change in IGFBP-3 SDS.

Safety analysis set and On-treatment are used to present the primary estimand for the primary objective and all other safety data.


 Date:
 24 June 2022
 Novo Nordisk

 Version:
 1.0

 Status:
 Final

 Page:
 13 of 24

## 4 Statistical Analyses

#### 4.1 General Considerations

Descriptive statistics will be performed as described in the sections 4.2 and 4.3.

#### 4.2 Primary Endpoint/Estimand Analysis

The primary endpoint number of adverse events will be used to support the primary objective of evaluating safety of once-weekly somapacitan during 26 weeks of treatment in children with SGA, TS, NS or ISS based on the primary estimand corresponding to the on-treatment data points set.

To support the primary estimand descriptive statistics (Number and percentage of participants who experienced adverse events, the number of events) will be derived in addition to the event rate per 100 patient years of exposure. The primary endpoint will be summarised for each indication, SGA,TS, NS or ISS. All adverse events with onset after the first administration of trial product and up until end of treatment or 14 days after last trial product administration, whichever comes first, will be included in the analysis. The adverse events will be summarised by MedDRA (Medical Dictionary for Regulatory Activities) system organ class and MedDRA preferred term. Adverse events with onset 14 days or more after last trial product administration will be reported in a separate listing.

#### 4.2.1 Definition of Endpoint

Number of adverse events (AEs) from baseline (week 0) to week 26.

#### 4.2.2 Main Analytical Approach

Safety analysis set and On-treatment are used to present the primary estimand for the primary objective.

#### 4.2.3 Sensitivity Analysis

Not applicable.

#### 4.2.4 Supplementary Analysis

Not applicable.

#### 4.3 Secondary Endpoints/Estimands Analysis

#### 4.3.1 Confirmatory Secondary Endpoints

Not applicable.

#### 4.3.2 Supportive Secondary Endpoints/Estimands

#### 4.3.2.1 Supportive secondary safety endpoints/estimands

The supportive secondary safety estimand regarding the incidence of AEs possibly or probably related to somapacitan from baseline up to week 26 of somapacitan treatment will be evaluated in a similar way as the primary endpoint including AEs possibly or probably related to somapacitan in the endpoint attribute.

The supportive secondary safety estimand regarding the incidence of AEs from baseline up to week

| Statistical Analysis Plan | | Date: | 24 June 2022 <b>Nove</b> | o Nordisk |
|---|---|---|---|---|
| · | CONFIDENTIAL | Status: | Final | |
| | | Page: | 14 of 24 | |

156 of somapacitan treatment will be evaluated in a similar way as the primary endpoint substituting 156 weeks for 26 weeks.

#### 4.3.2.2 Supportive secondary efficacy endpoints/estimands

#### Table 1 Supportive secondary efficacy endpoints

| Title | Time frame | Unit |
|---|---|---|
| Height velocity | From baseline (week 0) to visit 7 (week 26) | cm/year |
| Change in Height SDS | From baseline (week 0) to visit 7 (week 26) | Score <sup>a</sup> |
| Change in Height Velocity SDS | From baseline (week 0) to visit 7 (week 26) | Score <sup>a</sup> |
| Change in IGF-I SDS | From baseline (week 0) to visit 7 (week 26) | Score <sup>a</sup> |
| Change in IGFBP-3 SDS | From baseline (week 0) to visit 7 (week 26) | Score <sup>a</sup> |
| Weekly average somapacitan concentration $(C_{avg})$ based on population PK analysis | From baseline (week 0) to visit 7 (week 26) | ng/ml |

<sup>&</sup>lt;sup>a</sup>Positive score indicates that the value is closer to or above the reference population compared to baseline.

### Height velocity, Change in Height SDS and Change in Height Velocity SDS

The clinical question of interest for the supportive secondary efficacy endpoints Height velocity, Change in Height SDS and Change in Height Velocity SDS are: What is the mean Height velocity, Change in Height SDS or Change in Height Velocity SDS after 26 weeks of somapacitan treatment for each group of previously treated (yes/no) in the four populations (SGA, TS, NS or ISS) regardless of dose reduction due to IGF-I or AE, regardless of treatment discontinuation for any reason and regardless of initiation of ancillary therapy or medication with a special focus?

The supportive secondary estimands are defined for each of the four populations (SGA, TS, NS or ISS) with five attributes:

- The treatment condition of interest is defined as somapacitan treatment with or without ancillary therapy or medication with a special focus (treatment policy strategy).
- The population targeted by the clinical question: The treatment effect will be assessed separately for each group of previously treated (yes/no) in the four populations (SGA, TS, NS or ISS).
- Endpoints:
- Height velocity from baseline (week 0) to visit 7 (week 26)
- Change in Height SDS from baseline (week 0) to visit 7 (week 26)
- Change in Height Velocity SDS from baseline (week 0) to visit 7 (week 26)

Remaining intercurrent events: The 4 intercurrent events 'dose reduction due to IGF-I or AE', 'treatment discontinuation for any reason', 'initiation of ancillary therapy' and 'medication with a special focus', are all addressed by the treatment condition of interest attribute. There are no remaining intercurrent events.

• Population-level summary: Mean change

Rationale for estimands: The estimands assess the expected benefit a future population (SGA, TS, NS or ISS) can achieve if prescribed somapacitan. By not placing any restrictions on treatment adherence, these estimands aim to obtain a difference as close as possible to the one that can be expected in clinical practice, provided that the dose reduction, treatment adherence and use of ancillary therapy in the study reflects what would be seen in clinical practice.

| Statistical Analysis Plan | | Date: | 24 June 2022 | Novo Nordisk |
|---|---|---|---|---|
| • | CONFIDENTIAL | Status: | Status: Final | |
| | | Page: | 15 of 24 | |

The supportive secondary estimands will be evaluated based on all participants where both baseline and week 26 data are collected. To support the supportive secondary estimands SD, median, min and max values will also be derived for the supportive secondary endpoints.

#### Change in IGF-I SDS and Change in IGFBP-3 SDS

The clinical question of interest for the supportive secondary efficacy endpoints Change in IGF-I SDS and Change in IGFBP-3 SDS from baseline (week 0) to visit 7 (week 26) are: What is the mean change after 26 weeks of somapacitan treatment within each group of previously treated (yes/no) in the four populations (SGA, TS, NS or ISS) patients while on treatment regardless of dose reduction due to IGF-I or AE or medication with a special focus?

The supportive secondary estimands are defined for each of the four populations (SGA, TS, NS or ISS) with five attributes:

- The treatment condition of interest is defined as somapacitan regardless of dose reduction or medication with a special focus.
- The population targeted by the clinical question: The treatment effect will be assessed separately for each group of previously treated (yes/no) in the four populations (SGA, TS, NS or ISS)
- Endpoints:
  - o Change in IGF-I SDS from baseline week 0 to week 26
  - o Change in IGFBP-3 SDS from baseline week 0 to week 26
- Remaining intercurrent events:
  - Treatment discontinuation for any reason: Participant's data will be included up to 14 days after treatment discontinuation. Data collected 14 days after the intercurrent event will be regarded as not relevant for the estimation of the treatment effect.
  - o Initiation of medication with a special focus: Addressed by the treatment condition of interest attribute.
  - O Dose reduction due to IGF-I or AE: Addressed by the treatment condition of interest attribute. There are no remaining intercurrent events.
- Population-level summary: Mean change

Rationale for estimand: The supportive secondary estimand assesses the expected benefit a future population (SGA, TS, NS or ISS) can achieve if prescribed somapacitan if no treatment discontinuation had occurred.

The supportive secondary estimands will be evaluated based on all participants where both baseline and week 26 data are collected. To support the supportive secondary estimands SD, median, min and max values will also be derived for the supportive secondary endpoints.

FAS and In-study are used to estimate the supportive secondary efficacy estimands for Height velocity, Change in Height SDS and Change in Height Velocity SDS.

FAS and On-treatment are used to present the supportive secondary efficacy estimands for Change in IGF-I SDS and Change in IGFBP-3 SDS.

### Pharmacokinetic and/or pharmacodynamic modelling

Pharmacokinetic (PK) and pharmacodynamic (PD) modelling based on the somapacitan concentration and IGF-I data from the study will be performed.

| Study ID: NN8640-4469 CONFIDENTIAL S | Date: 24 June 2022 Version: 1.0 Status: Final | Novo Nordisk |
|---|---|---|
|---|---|---|

The objective of the PK/PD modelling analysis is to characterise the weekly PK/PD profile, weekly average exposure (C<sub>avg</sub>) and weekly IGF-I average levels following somapacitan treatment in SGA, TS, NS and ISS.

A more technical and detailed elaboration of the PK/PD modelling will be given in a modelling analysis plan (MAP), which will be prepared prior to database lock. Weekly average exposure (C<sub>avg</sub>) based on population PK/PD modelling will be reported as a secondary endpoint. Other PK/PD modelling results will be reported in a separate modelling report, which will not be part of the CSR. The individual somapacitan concentration data will be tabulated in the bioanalytical report.

#### 4.4 Exploratory Endpoints Analysis

Not applicable.

#### 4.5 Other Safety Analysis

### Safety laboratory assessments

Safety laboratory assessments (biochemistry, haematology, glucose metabolism, coagulation parameters (NS), and lipids) will be summarised by time of assessment for each indication, SGA, TS, NS or ISS. All abnormal values will be listed.

#### Vital signs

Vital signs (electrocardiogram, transthoracic electrocardiogram (TS, NS)) will be summarised by time of assessment for each indication, SGA, TS, NS or ISS. The investigator's evaluation of vital signs will be tabulated by time of assessment for each indication, SGA, TS, NS or ISS.

#### **Antibodies**

For confirmed anti-somapacitan antibody positive samples, the anti-somapacitan positive crossreactivity to hGH antibodies and in vitro neutralising effect will be tabulated by time of assessment for each indication, SGA, TS, NS or ISS.

#### 4.5.1 Extent of Exposure

Not applicable.

#### 4.5.2 Adverse Events

Adverse events will be displayed as per the primary and secondary endpoints.

#### 4.5.3 Additional Safety Assessments

Not applicable.

#### 4.6 Other Analysis

### 4.6.1 Other parameters


Date: 24 June 2022 Novo Nordisk Version: 1.0 Status: Final 17 of 24 Page:

#### Table 2 Overview of other parameters

| Title | Time frame | Unit |
|---|---|---|
| Child treatment burden measure: GH-INJ-CTB-Physical <sup>e</sup> | Visit 5 | Score <sup>a</sup> |
| Child treatment burden measure: GH-INJ-CTB-Emotional Well-being <sup>e</sup> | Visit 5 | Score <sup>a</sup> |
| Child treatment burden measure: GH-INJ-CTB-Interference <sup>e</sup> | Visit 5 | Score <sup>a</sup> |
| Child treatment burden measure: GH-INJ-CTB-Overall treatment burden <sup>e</sup> | Visit 5 | Score <sup>a</sup> |
| Patient Preference: GH-PPQ-Childe | Visit 5 | Categorical response |
| Near adult height (NAH) | 18 months prior to screening to visit 18 (week 156) | Yes/No |
| Change in height SDS at the visit when NAH is reached | From baseline (week 0) to the visit NAH is reached | Score <sup>b</sup> |
| Midparental target height (MPH) | Screening (visit 1) | cm |
| MPH SDS | Screening (visit 1) | Score <sup>c</sup> |
| Index of genetic height potential | From baseline (week 0) to the visit NAH is reached | Score <sup>d</sup> |
| Change in interventricular Septum end diastole (IVSed) SDS | From baseline (week 0) to visit 7 (week 26) | Score <sup>b</sup> |
| Change in left ventricle posterior wall end diastole (LVPWed) SDS | From baseline (week 0) to visit 7 (week 26) | Score <sup>b</sup> |
| Change in left ventricle inner dimension end diastole (LVIDed) SDS | From baseline (week 0) to visit 7 (week 26) | Score <sup>b</sup> |
| Change in left ventricle inner dimension end systole (LVIDes) SDS | From baseline (week 0) to visit 7 (week 26) | Score <sup>b</sup> |
| Change in sitting height/height (SH/H) | From baseline (week 0) to visit 7 (week 26) | Ratio |
| Change in sitting height/height SDS (SH/H SDS) | From baseline (week 0) to visit 7 (week 26) | Ratio |
| Change in bone age/chronological age | From screening (visit 1) to visit 9 (week 52) | Ratio |

<sup>&</sup>lt;sup>a</sup>Negative score indicates that treatment burden is less compared to baseline.

Height Velocity at visit 9 (week 52), Change in Height SDS from baseline (week 0) to visit 9 (week 52), Change in Height Velocity SDS from baseline (week 0) to visit 9 (week 52), Change in IGF-1 SDS from baseline (week 0) to visit 9 (week 52) and Change in IGFBP-3 SDS from baseline (week 0) to visit 9 (week 52) will derived as parameters in the same way as the corresponding secondary endpoints at visit 7 (week 26).

The parameters will be summarised for relevant indications, SGA, TS, NS or ISS.

#### 4.6.2 **Subgroup Analysis**

Not applicable.

#### 4.7 **Interim Analysis**

Not applicable.

<sup>&</sup>lt;sup>b</sup>Positive score indicates that the value is closer to or above the reference population compared to baseline.

<sup>&</sup>lt;sup>c</sup>Negative values indicate that the values are lower than the reference population.

<sup>&</sup>lt;sup>d</sup>Negative values indicate that the NAH is below the genetic height potential.

<sup>&</sup>lt;sup>e</sup>Only to be collected from participants switching to somapacitan from daily GH treatment.

Statistical Analysis Plan
Study ID: NN8640-4469


Date: 24 June 2022 Version: 1.0
Status: Final 

## 4.8 Changes to Protocol-planned Analysis

There are no changes to the protocol-planned analysis.

| Statistical Analysis Plan |
|---------------------------|
| Study ID: NN8640-4469 |


Date: 24 June 2022 Novo Nordisk
Version: 1.0
Status: Final


# 5 Sample size determination

No formal sample size calculation was performed in the four populations (SGA, TS, NS or ISS). The number of participants reflects what is expected feasible to enroll to provide adequate safety information in each indication.

Children above or equal to 10.0 years (girls with SGA, TS, NS and ISS) or 11.0 years (boys with SGA, NS and ISS) and below 18.0 years are not included in the pivotal study NN8640-4467. Based on a recommendation from the FDA, this age group will be investigated in study NN8640-4469.

Up to 50 participants are planned to be enrolled in this study. In total, at least 10 participants in each indication are planned to complete the study, as outlined below:

- **SGA:** Ten (10) female and male participants equal to or above 10.0 and 11.0 years, respectively, and below 18.0 years at screening.
- **TS:** Ten (10) female participants equal to or above 10.0 years and below 18.0 years at screening.
- NS: Ten (10) female and male participants equal to or above 10.0 and 11.0 years, respectively, and below 18.0 years at screening.
- **ISS:** Ten (10) female and male participants equal to or above 10.0 and 11.0 years, respectively, and below 18.0 years at screening.


24 June 2022 Novo Nordisk Date: Version: 1.0 Status: Final 

#### **Supporting Documentation** 6

#### Appendix 1: Definition and calculation of endpoints, assessments and derivations 6.1

| Type | Title | Time frame | Unit | Details |
|---|---|---|---|---|
| Supportive<br>secondary<br>efficacy<br>endpoint | Height velocity | From baseline (week 0) to visit 7 (week 26). | cm/year | Derived as: HV at week 26 = (height at 26 weeks visit – height at baseline)/(time from baseline to 26 weeks visit in years). |
| Supportive<br>secondary<br>efficacy<br>endpoint | Change in Height<br>SDS | From baseline (week 0) to visit 7 (week 26). | Score <sup>b</sup> | Derived as the Height SDS value at baseline week 0 subtracted from the Height SDS value at week 26 (visit 7). Height SDS is derived as: $ \frac{\left(\frac{\text{Height}_i}{\text{population median}}\right)^{\text{Skewness}} - 1}{\text{Skewness}} \times \text{population SD} $ where i indicates the visit. The population median and standard deviation are the ones corresponding to the age at visit i. The population median and standard deviation and skewness are based on reference data. $^1$ |
| Supportive<br>secondary<br>efficacy<br>endpoint | Change in Height<br>Velocity SDS | From baseline (week 0) to visit 7 (week 26). | Score <sup>b</sup> | Derived as the Height Velocity SDS value at baseline week 0 subtracted from the Height Velocity SDS value at week 26 (visit 7). Height Velocity SDS is derived as: $HVSDS_i = \frac{HV_i - populationmeanHV}{populationSD}$ where i indicates the visit. The population mean and standard deviation corresponding to the age at visit i. The population mean and standard deviation are based on reference data. $\frac{1.2}{1.2}$ |
| Supportive<br>secondary<br>efficacy<br>endpoint | Change in IGF-I<br>SDS | From baseline (week 0) to visit 7 (week 26). | Score <sup>b</sup> | Derived as the IGF-I SDS value at baseline week 0 subtracted from the IGF-I SDS value at week 26 (visit 7). IGF-I SDS is derived as: $IGF-I \ SDS_i = \frac{\left(\frac{IGF-I_i}{population\ median}\right)^{Skewness}-1}{Skewness\ *\ population\ SD}$ where i indicates the visit. The population median and standard deviation are the ones corresponding to the age at visit i. The population median and standard deviation and skewness are based on reference data. $\frac{3}{2}$ |
| Supportive<br>secondary<br>efficacy<br>endpoint | Change in<br>IGFBP-3 SDS | From baseline (week 0) to visit 7 (week 26). | Score <sup>b</sup> | Derived as the IGFBP-3 SDS value at baseline week 0 subtracted from IGFBP-3 SDS value at week 26 (visit 7). IGFBP-3 SDS is derived as: $IGFBP-3 SDS_{i} = \frac{\left(\frac{IGFBP-3_{i}}{population\ median}\right)^{Skewness}-1}{Skewness\ *\ population\ SD}$ where i indicates the visit. The population median and standard deviation are the ones corresponding to the |


Date: Version: Status: Final 

24 June 2022 | Novo Nordisk 1.0

| | 1 | 1 | 1 | |
|---|---|---|---|---|
| | | | | age at visit i. The population median and standard |
| | | | | deviation and skewness are based on reference data. <sup>4</sup> |
| Other parameter | Child treatment | Visit 5 | Scorea | GH-INJ-CTB-Physical score at week 13 (visit 5). |
| • | burden<br>measure: GH-<br>INJ-CTB-<br>Physical <sup>e</sup> | | | GH-INJ-CTB – Physical score is derived as the sum of the 4 items (0=Not at all, 1=A little, 2=Some, 3=A lot, 4=Extreme) normalised to a 0-100-point scale as: |
| Other parameter | Child treatment | Visit 5 | Score <sup>a</sup> | Physical (question 1-4): (Sum/16)*100 GH-INJ-CTB-Emotional Well-being score at week 13 (visit 5). |
| | burden<br>measure: GH-<br>INJ-CTB-<br>Emotional<br>Well-being <sup>e</sup> | | | GH-INJ-CTB – Emotional Well-being score is derived as the sum of the 4 items (0=Not at all, 1=A little, 2=Some, 3=A lot, 4=Extreme) normalised to a 0-100-point scale as: |
| Other | Child | Visit 5 | Score <sup>a</sup> | Emotional Well-being (question 5-10): (Sum/24)*100 GH-INJ-CTB-Interference score at week 13 (visit 5). |
| parameter | treatment<br>burden<br>measure: GH-<br>INJ-CTB-<br>Interference <sup>c</sup> | | | GH-INJ-CTB – Interference score is derived as the sum of the 4 items (0=Not at all, 1=A little, 2=Some, 3=A lot, 4=Extreme) normalised to a 0-100-point scale as: Interference: (question 11-14): (Sum/16)*100 |
| Other parameter | Child<br>treatment<br>burden | Visit 5 | Scorea | GH-INJ-CTB-Overall treatment burden score at week 13 (visit 5). |
| | measure: GH-<br>INJ-CTB-Overall<br>treatment<br>burden <sup>c</sup> | | | GH-INJ-CTB – Overall treatment burden score is derived as the mean of the GH-INJ-CTB – Physical score, GH-INJ-CTB - Emotional Well-being score and GH-INJ-CTB – Interference score. |
| Other parameter | Patient Preference: GH-PPQ-Childe | Visit 5 | Categorical response | Patient Preference GH-PPQ-Child at week 13 (visit 5) (Previous treatment, Current treatment, No preference). |
| Other<br>parameter | Near adult<br>height (NAH) | 18 months<br>prior to<br>screening to<br>visit 18<br>(week 156) | Yes/No | Near adult height (NAH) will be derived. NAH is defined as HV < 2 cm/year calculated over a period of at least 9 months, males have reached a bone age of ≥16 years and females has reached a bone age of ≥14 years. If bone age is not available, then males have reached a chronological age of ≥17 years and females have reached a chronological age of ≥15 years. Historical height measurements collected at screening will be included in the derivation. |
| Other<br>parameter | Change in<br>height SDS at<br>the visit when<br>NAH is reached | From baseline (week 0) to the visit NAH is reached | Scoreb | Derived as the Height SDS value at baseline week 0 subtracted from the Height SDS value at the visit where NAH is reached. |
| Other<br>parameter | Midparental<br>target height<br>(MPH) | Screening (visit 1) | cm | Derived as: Girls TH: (mother's height + father's height-13)/2. <sup>5</sup> Boys TH: (mother's height + 13 + father's height)/2. <sup>5</sup> |
| Other<br>parameter | MPH SDS | Screening (visit 1) | Score <sup>c</sup> | MPH SDS is derived as: MPH SDS = Fathers height SDS + mothers height SDS 2 |

| Statistical Analysis Plan | | Date: | 24 June 2022 | Novo Nordisk |
|---|---|---|---|---|
| · | CUNFIDENTIAL | G | Tr: 1 | |

Status:

Final

 Where parental height SDS is derived as: Parental height SDS =  $\frac{\text{Height - population mean}}{\text{nonulation SD}}$ The population mean and standard deviation comes from reference data.6 Other Derived as NAH SDS - MPH SDS Index of From Scored baseline parameter genetic height potential (week 0) to the visit NAH is reached Scoreb Derived as the IVSed SDS value at baseline week 0 Other Change in From parameter interventricular baseline subtracted from IVSed SDS value at week 26 (visit 7) Septum end (week 0) to for Turner syndrome. diastole visit 7 (week (IVSed) SDS IVSed SDS is derived as: 26) IVSed SDS<sub>i</sub>  $\underline{ln(IVSed\ SDS)_i - intercept + ln(Weight_i*slope)}$ where i indicates the visit. The intercept, slope and SD residuals are the ones corresponding to the age at visit i. The intercept, slope and SD residuals are based on reference data.<sup>7</sup> Other Change in left Score<sup>b</sup> Derived as the LVPWed SDS value at baseline week 0 From parameter ventricle baseline subtracted from LVPWed SDS value at week 26 (visit posterior wall (week 0) to 7) for Turner syndrome. end diastole visit 7 (week (LVPWed) LVPWed SDS is derived as: 26) SDS LVPWe SDS<sub>i</sub> ln(LVPWe SDS)<sub>i</sub> - intercept + ln(Weight<sub>i</sub> \* slope) SD residual where i indicates the visit. The intercept, slope and SD residuals are the ones corresponding to the age at visit i. The intercept, slope and SD residuals are based on reference data.<sup>7</sup> Scoreb Derived as the LVIDed SDS value at baseline week 0 Other Change in left From subtracted from LVIDed SDS value at week 26 (visit 7) parameter ventricle inner baseline dimension end (week 0) to for Turner syndrome. diastole visit 7 (week (LVIDed) SDS 26) LVIDed SDS is derived as: LVIDed SDS<sub>i</sub>  $ln(LVIDed SDS)_i - intercept + ln(Weight_i * slope)$ 

where i indicates the visit. The intercept, slope and SD residuals are the ones corresponding to the age at visit i. The intercept, slope and SD residuals are based on reference data. 7 Change in left Other Derived as the LVIDes SDS value at baseline week 0 From Scoreb ventricle inner baseline subtracted from LVIDes SDS value at week 26 (visit 7) parameter dimension end (week 0) to for Turner syndrome. visit 7 (week systole (LVIDes) SDS LVIDes SDS is derived as:

| | | | | |
|---|---|---|---|---|
| | | | | $LVIDes SDS_{i} \\ = \frac{\ln(LVIDes SDS)_{i} - intercept + \ln(Weight_{i} * slope)}{SD \text{ residual}}$ where i indicates the visit. The intercept, slope and SD residuals are the ones corresponding to the age at visit i. The intercept, slope and SD residuals are based on reference data. The intercept is the substant of the s |
| Other parameter | Change in sitting height/height (SH/H) | From baseline (week 0) to visit 7 (week 26) | Ratio | Derived as SH/H at baseline week 0 subtracted from SH/H at week 26 (visit 7) for <b>TS &amp; ISS</b> . |
| Other parameter | Change in<br>sitting<br>height/height<br>SDS (SH/H<br>SDS) | From baseline (week 0) to visit 7 (week 26) | Ratio | Derived as SH/H SDS at baseline week 0 subtracted from SH/H SDS at week 26 (visit 7) for <b>TS &amp; ISS</b> . SH/H SDS is derived as: |

Date:


Version:

Status:

24 June 2022 | Novo Nordisk

Skewness \* population SD

where i indicates the visit. The population median and standard deviation are the ones corresponding to the age

(visit 1) subtracted from the bone age/chronological age

The bone age/chronological age value at screening

value at week 52 (visit 9).

1.0

Final

From

screening

(visit 1) to

visit 9 (week

Statistical Analysis Plan

Study ID: NN8640-4469

Other

parameter

Change in

age/chronological

bone

age

Ratio

<sup>52)</sup> <sup>a</sup>Negative score indicates that treatment burden is less compared to baseline.

Positive score indicates that the value is closer to or above the reference population compared to baseline.

<sup>&</sup>lt;sup>c</sup>Negative values indicate that the values are lower than the reference population.

<sup>&</sup>lt;sup>d</sup>Negative values indicate that the NAH is below the genetic height potential.

<sup>&</sup>lt;sup>e</sup>Only to be collected from participants switching to somapacitan from daily GH treatment.

| Statistical Analysis Plan Study ID: NN8640-4469 CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 24 June 2022<br>1.0<br>Final<br>24 of 24 | Novo Nordisk |
|---|---|---|---|
|---|---|---|---|

### 7 References

1. Kuczmarski RJ. CDC growth Charts: United States. Advanced data from vital and health statistics. 2000.

- 2. Prader. Physical growth of Swiss children from birth to 20 years of age: first Zurich longitudinal study of growth and development. Helv Paediatr Acta Suppl. 52:1-1251989 1989.
- 3. Bidlingmaier M, Friedrich N, Rebecca T, Emeny JS, Wolthers OD, Roswall J, et al. Reference Intervals for Insulin-like Growth Factor-1 (IGF-I) From Birth to Senescence: Results From a Multicenter Study Using a New Automated Chemiluminescence IGF-I Immunoassay Conforming to Recent International Recommendations. J Clin Endocrinol Metab. 2014;99(5):1712-21.
- 4. Friedrich N, Wolthers OD, Arafat AM, Emeny RT, Spranger J, Roswall J, et al. Age- and sex-specific reference intervals across life span for insulin-like growth factor binding protein 3 (IGFBP-3) and the IGF-I to IGFBP-3 ratio measured by new automated chemiluminescence assays. J Clin Endocrinol Metab. 2014;99(5):1675-86.
- 5. Tanner JM, Goldstein H, Whitehouse RH. Standards for Children's Height at Age 2 to 9 years allowing for height of Parents. Arch Dis Child. 1970;45(244):819.
- 6. Cole TJ. Galton's midparent height revisited. Ann Hum Biol. 2000;27(4):401-5.
- 7. Overbeek LI, Kapusta L, Peer PG, de Korte CL, Thijssen JM, Daniels O. New reference values for echocardiographic dimensions of healthy Dutch children. Eur J Echocardiogr. 2006;7(2):113-21.